CLINICAL TRIAL: NCT02177175
Title: Carvedilol for the Prevention of Anthracycline/Anti-HER2 Therapy Associated Cardiotoxicity Among Women With HER2-Positive Breast Cancer Using Myocardial Strain Imaging for Early Risk Stratification
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-099
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: Carvedilol; Anthracycline; HER2; 14-099
MeSH Terms: conditions — Breast Neoplasms | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Carvedilol (Experimental): Treatment in both carvedilol and placebo groups will be systematically up-titrated at weeks 3, 6, and 9 (+/- 1 week) after randomization to a goal dose of 25mg twice daily.
  Interventions: Drug: Carvedilol
- placebo (Placebo Comparator): Treatment in both carvedilol and placebo groups will be systematically up-titrated at weeks 3, 6, and 9 (+/- 1 week) after randomization to a goal dose of 25mg twice daily.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Carvedilol
  Arms: Carvedilol
Other: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to find out the effects, good and/or bad, of a beta blocker (carvedilol) on heart function during treatment with anti-HER2 medication(s) including trastuzumab (Herceptin).

DETAILED DESCRIPTION:
This phase II placebo-controlled study will evaluate the effect of carvedilol, compared to placebo, on anthracycline/anti-HER2 therapy induced left ventricular dysfunction in patients with HER2-positive breast cancer who are receiving adjuvant or neoadjuvant therapy. All patients will undergo routine cardiac surveillance with 2D echocardiograms per standard of care at multiple time points which will align as closely as possible to the following: pre-anthracycline (baseline), pre-anti-HER2 therapy, and 3, 6, 9, and 12 months (+/- 4 weeks) after initiation of anti-HER2 therapy. In the case that standard of care echocardiograms are not done at these time points, either due to a delay in anti-cancer therapy or due to the patient's medical condition, the principal investigator will determine if the standard of care echocardiogram may be used in lieu of one of the time points listed. Additional speckle tracking strain analysis will be performed on these echocardiograms, and blood specimens will be drawn at several time points for biomarker analysis.

After completion of anthracycline treatment and prior to initiation of anti-HER2 therapy, 32 patients with abnormal myocardial strain, defined as global longitudinal strain < 19% or % change from baseline by > 11%, will be randomized in a 1:1 ratio to carvedilol versus placebo. Carvedilol will be administered twice daily for approximately 1 year OR until the end of anti-HER2 therapy, if it is discontinued prior to 1 year. Treatment in both carvedilol and placebo groups will be systematically up-titrated at weeks 3, 6, and 9 (+/- 1 week) after randomization to a goal dose of 25mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18 years
* Non-metastatic histologically confirmed primary invasive breast carcinoma
* Pathologically confirmed HER2-positive breast cancer
* Scheduled to receive anthracycline chemotherapy followed by anti-HER2 therapy at MSKCC
* Able and willing to provide informed consent
* Willing and able to comply with the requirements of the protocol
* Able to swallow capsules

For Aim 2, all patients must meet the following criteria:

* Meet all inclusion criteria above

  * LVEF > 50%
* Abnormal global longitudinal strain (<19%, or a % decrease of ≥ 11% from baseline) prior to initiation of planned anti-HER2 therapy
* Heart rate ≥ 50 beats per minute
* Sitting systolic blood pressure > 90 mmHg

Exclusion Criteria:

* Patients are to be excluded from randomization for Aim 2 of this study if they meet any of the following criteria:
* Current treatment with ACE-inhibitors or beta blockers
* Allergies or inability to tolerate beta blockers previously due to bradycardia, hypotension, or AV block.
* Known history of NCI CTCAE (Version 4.0) Grade ≥ 2 symptomatic CHF, myocardial infarction within 12 months prior to randomization, significant symptoms (Grade ≥ 3) relating to left ventricular dysfunction, significant (moderate or severe) valvular disease, or significant cardiac arrhythmia (Grade ≥ 3)
* Pre-menopausal women without a negative serum or urine pregnancy test within 4 weeks of starting treatment
* Enrollment in a therapeutic intervention trial in the Breast Medicine service

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Yu AF, Moore ZR, Moskowitz CS, Liu JE, Dang CT, Ramanathan L, Oeffinger KC, Steingart RM, Schmitt AM. Association of Circulating Cardiomyocyte Cell-Free DNA With Cancer Therapy-Related Cardiac Dysfunction in Patients Undergoing Treatment for ERBB2-Positive Breast Cancer. JAMA Cardiol. 2023 Jul 1;8(7):697-702. doi: 10.1001/jamacardio.2023.1229. PMID 37256614
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants were randomized to treatment. 71 participants were not randomized to treatment.
Groups:
- Carvedilol: Treatment in both carvedilol and placebo groups will be systematically up-titrated at weeks 3, 6, and 9 (+/- 1 week) after randomization to a goal dose of 25mg twice daily.
  Carvedilol
- Placebo: Treatment in both carvedilol and placebo groups will be systematically up-titrated at weeks 3, 6, and 9 (+/- 1 week) after randomization to a goal dose of 25mg twice daily.
  placebo
Period: Overall Study
Arm/Group | Carvedilol | Placebo
Started | 5 | 6
Completed | 4 | 6
Not Completed | 1 | 0
Not completed — stopped trastuzumab so was taken off study | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carvedilol | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Full Range); unit: years] | 45.6 [38 to 52] | 55.2 [38 to 65] | 50.8 [38 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change in LVEF at 3 Months
Description: Value at 3 months minus value at baseline
Time Frame: 3 months
Measure: Median (Full Range); unit: change in percent ejection fraction
Arm/Group | Carvedilol | Placebo
Number analyzed (Participants) | 5 | 6
change in percent ejection fraction | 1 [-3 to 6] | -5 [-12 to 0]

2. Primary Outcome: Maximum Change in LVEF at 6 Months
Description: Value at 6 months minus value at baseline
Time Frame: 6 months
Measure: Median (Full Range); unit: change in percent ejection fraction
Arm/Group | Carvedilol | Placebo
Number analyzed (Participants) | 5 | 6
change in percent ejection fraction | -2 [-7 to 1] | -5 [-7 to 4]

3. Primary Outcome: Maximum Change in LVEF at 9 Months
Description: Value at 9 months minus value at baseline
Time Frame: 9 months
Measure: Median (Full Range); unit: change in percent ejection fraction
Arm/Group | Carvedilol | Placebo
Number analyzed (Participants) | 5 | 6
change in percent ejection fraction | -3.5 [-4 to -3] | -5.5 [-13 to 4]

4. Primary Outcome: Maximum Change in LVEF at 12 Months
Description: Value at 12 months minus value at baseline
Time Frame: 12 months
Measure: Median (Full Range); unit: change in percent ejection fraction
Arm/Group | Carvedilol | Placebo
Number analyzed (Participants) | 5 | 6
change in percent ejection fraction | -2.5 [-4 to 1] | -2 [-13 to 4]

5. Secondary Outcome: Incidence of Abnormal LVEF at 12 Months
Description: The study is designed to detect an intergroup difference of absolute difference of 10 percentage points (simple difference) in the change in LVEF between the experimental and control group. Ten percent is the change in LVEF that is associated with differing degrees of left ventricular dysfunction, and long-term studies among non-cancer patients have shown that outcomes differ among groups of patients who have LVEF differing by 10%.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carvedilol | Placebo
Number analyzed (Participants) | 5 | 6
Participants
  Abnormal LVEF | 2 | 1
  Normal LVEF | 3 | 5

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Carvedilol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/6
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carvedilol (N=5) | Placebo (N=6)
Skin infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carvedilol (N=5) | Placebo (N=6)
Alanine aminotransferase increased (Investigations) | 3 | 1
Alkaline phosphatase increased (Investigations) | 4 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 6
Aspartate aminotransferase increased (Investigations) | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 2 | 2
White blood cell decreased (Investigations) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT02177175/Prot_SAP_000.pdf